CLINICAL TRIAL: NCT04689802
Title: To Identify Potential New Urine Marker Panel for Cancer Screening
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Professor, Chinese University of Hong Kong
Other Study IDs: CRE-2020.611
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Polyamines are naturally produced metabolites in our cells. There were some reports suggested the urinary levels of polyamines were altered in patients with different cancers. This study is to explore the use of urinary polyamine for the diagnosis of common cancers.

DETAILED DESCRIPTION:
Urine tests is a simple, non-invasive approach for cancer detection. One example of such cancer biomarkers are natural polyamines. Recently, there are also other reports on the use of polyamines in diagnosis of other cancers. In this larger scale study, with inclusion of subjects with different cancer types, to further assess the correlation urine polyamines and other urine metabolite markers for the diagnosis of different cancer types and investigate their role as a potential non-invasive marker for cancer detection and monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with age > 18 years old.
2. For cancer patients, a histological diagnosis of cancer is available.
3. For normal control, there is no diagnosis of cancer in the medical record.

Exclusion Criteria:

1. Patient with recent urinary tract infection within 6 weeks prior to urine collection.
2. Patient with recent urethral instrumentation, such as Foley catheter insertion, cystoscopy etc, within 6 weeks prior to urine collection.
3. Patient refused or unable to provide consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 2000 patients who has diagnosis of various cancers, and another 500 patients with no history of cancer will be recruited for the study. The sample size is based on the projected number of patients that can be recruited during the proposed study period.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of cancer detection by urine polyamines | 1 month after surgery
  Urine samples will be prepared and analyzed by ultra-high-performance liquid chromatography coupled with triple quadrupole mass spectrometer (UPLC-MS/MS). Receiver operating characteristics (ROC) curve for overall and individual cancer diagnosis will be performed.pathological result will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhang DZ, Lau KM, Chan ES, Wang G, Szeto CC, Wong K, Choy RK, Ng CF. Cell-free urinary microRNA-99a and microRNA-125b are diagnostic markers for the non-invasive screening of bladder cancer. PLoS One. 2014 Jul 11;9(7):e100793. doi: 10.1371/journal.pone.0100793. eCollection 2014. PMID 25014919
- [Background] Cheng THT, Jiang P, Teoh JYC, Heung MMS, Tam JCW, Sun X, Lee WS, Ni M, Chan RCK, Ng CF, Chan KCA, Chiu RWK, Lo YMD. Noninvasive Detection of Bladder Cancer by Shallow-Depth Genome-Wide Bisulfite Sequencing of Urinary Cell-Free DNA for Methylation and Copy Number Profiling. Clin Chem. 2019 Jul;65(7):927-936. doi: 10.1373/clinchem.2018.301341. Epub 2019 Apr 15. PMID 30988170
- [Background] Russell DH. Increased polyamine concentrations in the urine of human cancer patients. Nat New Biol. 1971 Sep 29;233(39):144-5. doi: 10.1038/newbio233144a0. No abstract available. PMID 5286749
- [Background] Lee SH, Yang YJ, Kim KM, Chung BC. Altered urinary profiles of polyamines and endogenous steroids in patients with benign cervical disease and cervical cancer. Cancer Lett. 2003 Nov 25;201(2):121-31. doi: 10.1016/s0304-3835(03)00014-4. PMID 14607325
- [Background] Loser C, Folsch UR, Paprotny C, Creutzfeldt W. Polyamines in colorectal cancer. Evaluation of polyamine concentrations in the colon tissue, serum, and urine of 50 patients with colorectal cancer. Cancer. 1990 Feb 15;65(4):958-66. doi: 10.1002/1097-0142(19900215)65:43.0.co;2-z. PMID 2297664
- [Background] Leveque J, Foucher F, Bansard JY, Havouis R, Grall JY, Moulinoux JP. Polyamine profiles in tumor, normal tissue of the homologous breast, blood, and urine of breast cancer sufferers. Breast Cancer Res Treat. 2000 Mar;60(2):99-105. doi: 10.1023/a:1006319818530. PMID 10845272
- [Background] Tsoi TH, Chan CF, Chan WL, Chiu KF, Wong WT, Ng CF, Wong KL. Urinary Polyamines: A Pilot Study on Their Roles as Prostate Cancer Detection Biomarkers. PLoS One. 2016 Sep 6;11(9):e0162217. doi: 10.1371/journal.pone.0162217. eCollection 2016. PMID 27598335
- [Background] Deng L, Ismond K, Liu Z, Constable J, Wang H, Alatise OI, Weiser MR, Kingham TP, Chang D. Urinary Metabolomics to Identify a Unique Biomarker Panel for Detecting Colorectal Cancer: A Multicenter Study. Cancer Epidemiol Biomarkers Prev. 2019 Aug;28(8):1283-1291. doi: 10.1158/1055-9965.EPI-18-1291. Epub 2019 May 31. PMID 31151939
- See also: Hong Kong Cancer Registry 2018. — https://www3.ha.org.hk/cancereg/pdf/overview/Overview%20of%20HK%20Cancer%20Stat%202018.pdf